CLINICAL TRIAL: NCT06700655
Title: A Clinical Study on Co-transplantation of Autologous Limbal Stem Cells and Corneal Stromal Stem Cells to Repair Corneal Injury: an Open-label, Randomized Clinical Trial
Brief Title: A Clinical Study on Co-transplantation of Autologous Limbal Stem Cells and Corneal Stromal Stem Cells to Repair Corneal Injury
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021GXB01-4
Record Dates: First submitted 2024-11-17; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Limbal Stem Cells Deficiency
Keywords: Limbal stem cell; Limbal stem cells deficiency; Corneal stromal stem cells; Corneal transplantation
MeSH Terms: interventions — Corneal Transplantation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cornea limbal stem cell transplantation group (Experimental): The corneal limbal tissue (2mm x 5mm) was harvested from the patient's healthy eye, and ex vivo amplification was performed to obtain an adequate quantity of transplantable corneal limbal stem cells The patient was followed up and re-examined for 2 years postoperatively.
  Interventions: Biological: Cornea limbal stem cell transplantation group
- Cornea limbal stem cell transplantation combined corneal stromal stem cell group (Experimental): The corneal limbal tissue (2mm x 5mm) was harvested from the patient's healthy eye, and ex vivo amplification was performed to obtain an adequate quantity of transplantable corneal limbal stem cells and corneal stromal stem cells. The patient was followed up and re-examined for 2 years postoperatively.
  Interventions: Biological: Cornea limbal stem cell transplantation combined corneal stromal stem cell group
- Corneal transplantation group (Active Comparator): The patient awaited allogeneic corneal donation and underwent corneal transplantation surgery. Postoperatively, the patient was followed up and re-examined for 2 years.
  Interventions: Procedure: Corneal transplantation

INTERVENTIONS:
Biological: Cornea limbal stem cell transplantation group — The corneal limbal tissue (2mm x 5mm) was harvested from the patient's healthy eye, and ex vivo amplification was performed to obtain an adequate quantity of transplantable corneal limbal stem cells.
  Arms: Cornea limbal stem cell transplantation group
Procedure: Corneal transplantation — The patient awaited allogeneic corneal donation and underwent corneal transplantation surgery.
  Arms: Corneal transplantation group
Biological: Cornea limbal stem cell transplantation combined corneal stromal stem cell group — The corneal limbal tissue (2mm x 5mm) was harvested from the patient's healthy eye, and ex vivo amplification was performed to obtain an adequate quantity of transplantable corneal limbal stem cells and corneal stromal stem cells.
  Arms: Cornea limbal stem cell transplantation combined corneal stromal stem cell group

SUMMARY:
This study aims to: 1) verify the feasibility of treating limbal stem cell deficiency (LSCD) caused by chemical injury with autologous limbal stem cell transplantation combined with corneal stromal stem cell transplantation; 2) evaluate the corneal healing patterns following autologous stem cell transplantation; and 3) establish a clinical intervention protocol based on autologous corneal stem cell transplantation. Sixty cases of single-eye LSCD were included.

DETAILED DESCRIPTION:
Limbal Stem Cells (LSCs) are the sole source of corneal epithelial self-renewal and play a critical role in maintaining corneal transparency. Chemical or physical injury to the eye and inflammation can lead to limbal stem cell deficiency (LSCD), accompanied by a series of pathological changes, such as irreversible fibrosis of corneal stromal cells and neovascularization, ultimately resulting in blindness. The fundamental solution for such diseases is the replenishment of LSCs to reconstruct a functional cornea. However, traditional treatment methods, such as corneal transplantation, face bottlenecks, including a severe shortage of corneal donors and the risk of immune rejection. Additionally, donor corneas do not contain LSCs, making it impossible to reconstruct the patient's limbal region, resulting in poor long-term efficacy.

In 2015, autologous LSCs were approved by the European Union as a commercial stem cell product for treating patients with chemically induced LSCD. However, LSCD patients are often accompanied by damage to the corneal stroma; while LSC transplantation can restore the limbal region and corneal epithelium, it cannot repair stromal opacities. Research indicates that transplantation of corneal stromal stem cells can reconstruct organized collagen structures and restore stromal transparency. Over the past decade, clinical studies using LSCs and corneal stromal stem cells to treat LSCD patients have been conducted in multiple countries, demonstrating the safety and efficacy of these stem cell therapies for corneal blindness.

Based on these findings above, the investigators have established a serum-free, carrier-free culture system that enables efficient and uniform in vitro expansion of functional LSCs and corneal stromal stem cells. By obtaining a 2 x 5 mm limbal tissue sample from the healthy eye of the patient, the investigators can acquire a sufficient number of cells for transplantation. Preclinical studies have confirmed that the expanded cells are effective and safe for treating LSCD animal models. This study aims to use autologous LSCs combined with corneal stromal stem cell transplantation to treat patients with unilateral LSCD, restoring their corneal transparency and visual function. This approach provides a novel treatment method for patients and promotes the application of stem cell regenerative medicine for the treatment of corneal blindness in China.

ELIGIBILITY:
Inclusion Criteria:

* Chemical injury from acid or alkali exposure
* Extensive limbal stem cell deficiency (greater than 180 degrees), with corneal stromal opacity not exceeding a depth of 250 μm
* Corneal epithelial conjunctivalization and fibrosis, with neovascularization extending into more than half of the quadrants
* Unilateral ocular involvement, with normal limbal stem cell function in the contralateral healthy eye
* No significant improvement in ocular surface signs and symptoms after pharmacological or surgical interventions, stable for over three months

Exclusion Criteria:

* Bilateral corneal stem cell deficiency, such as in Stevens-Johnson syndrome, ocular cicatricial pemphigoid, or congenital aniridia
* Subclinical limbal stem cell deficiency in the contralateral eye
* Signs of corneal endothelial decompensation, such as corneal bullae or corneal edema
* Presence of infectious inflammation on the ocular surface
* Severe dry eye
* Eyelid abnormalities requiring corrective surgery to restore normal anatomical structure
* Presence of chronic dacryocystitis, cataracts, uveitis, diabetic retinopathy, retinal detachment, or other ocular diseases
* Patients who have undergone cataract surgery or other intraocular procedures
* Glaucoma patients requiring long-term topical ocular medications
* History of corneal perforation in the affected eye
* Severe primary cardiovascular, hepatic, renal, endocrine, or hematologic disorders, diabetes, or immune deficiency in the medical history
* Pregnant or lactating women
* Positive screening for infectious diseases (HIV, HBV, HTLV, EBV, CMV, or syphilis)
* Other vision-impairing diseases present
* Allergy to bovine serum products
* History of multiple drug allergies or hypersensitive constitution
* Concurrent participation in other drug clinical trials
* History of mental health disorders affecting the ability to comply with study requirements
* Judged unsuitable for participation by the investigator

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Vision | [set the tissue sampling date at the begin] Enrollment, before the transplantation, First follow-up (Day 32), Second follow-up (Day 48), Third follow-up (Day 108), Fourth follow-up (6 months), Fifth follow-up (1 year), Sixth follow-up (2 years)
  The patient should initially be positioned 5 meters from the visual acuity chart in a well-lit environment. Each eye is tested separately (the non-tested eye should be completely covered with an eye patch without applying pressure on the eyeball). During the test, the patient first views the largest line on the chart. If they can identify it, they proceed from top to bottom, viewing progressively smaller lines until the smallest identifiable line is determined. The patient should not spend more than 5 seconds reading each character.

SECONDARY OUTCOMES:
Efficacy Scoring | [set the corneal limbal tissue sampling date at the begin] First follow-up (Day 32), Second follow-up (Day 48), Third follow-up (Day 108), Fourth follow-up (6 months), Fifth follow-up (1 year), Sixth follow-up (2 years)
  The efficacy of cell transplantation will be evaluated based on corneal epithelial defect, area of leukoplakia, transparency, neovascularization, and corneal edema.
Ocular adverse event evaluation | [set the corneal limbal tissue sampling date at the begin] before the transplantation, First follow-up (Day 32), Second follow-up (Day 48), Third follow-up (Day 108), Fourth follow-up (6 months), Fifth follow-up (1 year), Sixth follow-up (2 years)
  The transplantation area for the cells is the ocular surface, so the primary measure of safety will focus on post-transplant ocular symptoms. These include eye irritation symptoms, conjunctival hyperemia, corneal surface edema, and anterior chamber flare. Adverse events are defined as follows: eye irritation symptoms scoring ≥1, conjunctival hyperemia scoring ≥2, corneal surface edema scoring ≥2, anterior chamber flare scoring ≥2, or a total score of 7 or above.
  The healthy eye requires postoperative observation, and if infection or delayed healing occurs after tissue sampling, treatment will be necessary.
ophthalmic examination（slit-lamp） | [set the tissue sampling date at the begin] Enrollment, before the transplantation, First follow-up (Day 32), Second follow-up (Day 48), Third follow-up (Day 108), Fourth follow-up (6 months), Fifth follow-up (1 year), Sixth follow-up (2 years)
  including cornea, conjunctiva, lens, vitreous body and retina. Score each indicator from 0 to 3 based on the standards in the table, and then calculate the final score.
cornea confocal | [set the tissue sampling date at the begin] Enrollment, before the transplantation, Second follow-up (Day 48), Third follow-up (Day 108), Fourth follow-up (6 months), Fifth follow-up (1 year), Sixth follow-up (2 years)
  Corneal microscopic structure examination. Observe whether the morphology of each layer of the cornea is normal.
corneal topography | [set the tissue sampling date at the begin] Enrollment, before the transplantation, First follow-up (Day 32), Second follow-up (Day 48), Third follow-up (Day 108), Fourth follow-up (6 months), Fifth follow-up (1 year), Sixth follow-up (2 years)
  Analyze the morphology and curvature characteristics of the entire corneal surface.
Optical Coherence Tomography | [set the tissue sampling date at the begin] Enrollment, before the transplantation, First follow-up (Day 32), Second follow-up (Day 48), Third follow-up (Day 108), Fourth follow-up (6 months), Fifth follow-up (1 year), Sixth follow-up (2 years)
  Observe the depth of corneal lesions to assess the condition and treatment efficacy.
anterior segment photography | [set the tissue sampling date at the begin] Enrollment, before the transplantation, First follow-up (Day 32), Second follow-up (Day 48), Third follow-up (Day 108), Fourth follow-up (6 months), Fifth follow-up (1 year), Sixth follow-up (2 years)
  record the statement of ocular surface
VFQ-25 questionnaire | [set the tissue sampling date at the begin] Enrollment, before the transplantation, Second follow-up (Day 48), Third follow-up (Day 108), Fourth follow-up (6 months), Fifth follow-up (1 year), Sixth follow-up (2 years)
  The VFQ-25 (Visual Function Questionnaire-25) is a widely used tool to assess the health-related quality of life related to visual function. It consists of 25 questions to evaluate how vision affects daily activities, emotional well-being, and social interactions. The questionnaire covers several domains: general vision, near and distance vision, social functioning, role difficulties, mental health, and driving. It is often used in clinical settings to track the progression of eye diseases, evaluate treatment outcomes, or compare the quality of life between different patient groups. A higher score indicates better visual function and quality of life, meaning the patient experiences fewer difficulties and less impairment in daily activities due to vision problems. Therefore, higher scores are better in this context.

OTHER OUTCOMES:
Lung Condition | [set the tissue sampling date at the begin] Enrollment, Sixth follow-up (2 years)
  Evaluate lung conditions using a chest X-ray to rule out pulmonary nodules or other abnormalities. The specific findings are based on the hospital's chest X-ray report. A physician will determine their clinical significance if abnormalities are detected, considering factors such as correlation with the patient's medical history or whether the findings indicate an old lesion or non-pathological changes.
Cardiac Function | [set the tissue sampling date at the begin] Enrollment, Sixth follow-up (2 years)
  Evaluate myocardial function through electrocardiography (ECG) and X-ray, focusing on T-wave morphology, QT interval duration, and ST segment changes. Specific findings are based on the hospital's ECG report. The cardiac silhouette should also be assessed for signs of heart failure or pericardial effusion in X-ray. A physician will determine their clinical significance if abnormalities are detected, considering factors such as correlation with the patient's medical history or whether the findings indicate an old lesion or non-pathological variation.
Number of participants with abnormal hematologic parameters as assessed by standard criteria (the normal scale on the report) | [set the tissue sampling date at the begin] Enrollment, before the transplantation, Second follow-up (Day 48), Third follow-up (Day 108), Fifth follow-up (1 year), Sixth follow-up (2 years)
  Under fasting conditions, conduct blood tests for complete blood count (CBC), blood biochemistry, coagulation function, pregnancy test (for female participants), and infectious disease screening. Results are evaluated against the normal reference ranges provided in the lab report. If abnormalities are detected, a physician determines their clinical significance. Hematologic testing aims to identify potential systemic adverse events, such as rejection or infection (e.g., elevated white blood cell count), and assess for infectious diseases (e.g., HIV, hepatitis B, syphilis).
urine test | [set the tissue sampling date at the begin] Enrollment, First follow-up (Day 32), Fifth follow-up (1 year), Sixth follow-up (2 years)
  Urinalysis. The results are assessed against the normal reference ranges provided in the lab report. If abnormalities are identified, a physician will determine their clinical significance.
Head abnormalities in general physical condition as assessed by clinical examination | [set the tissue sampling date at the begin] Enrollment, First follow-up (Day 32), Fifth follow-up (1 year), Sixth follow-up (2 years)
  The examination is conducted according to the standards of the "Diagnostic Medicine (10th Edition, People's Medical Publishing House)".
  The head examination focuses on assessing the shape, symmetry, and condition of the scalp and facial features. Inspect for any deformities, scars, or abnormalities in the skull. Palpate for tenderness or masses, and observe for signs of trauma. The eyes should be examined for proper alignment, pupil size, and responsiveness. Check for conjunctival redness, discharge, or abnormalities. Inspect the nose for any deformities or discharge, and assess nasal patency. The ears should be examined for signs of infection, discharge, or abnormalities in shape and symmetry.
Neck abnormalities in general physical condition as assessed by clinical examination | [set the tissue sampling date at the begin] Enrollment, First follow-up (Day 32), Fifth follow-up (1 year), Sixth follow-up (2 years)
  The examination is conducted according to the standards of the "Diagnostic Medicine (10th Edition, People's Medical Publishing House)".
  The neck examination includes assessing the skin for any visible abnormalities such as scars or lumps. Palpate the neck for tenderness, masses, or enlarged lymph nodes. Examine the thyroid gland for enlargement, tenderness, or nodules. Assess the range of motion in the neck, and check for signs of pain, stiffness, or abnormal movement. Additionally, auscultate for any abnormal sounds, such as carotid bruits, that may indicate vascular abnormalities.
Lymph Node abnormalities in general physical condition as assessed by clinical examination | [set the tissue sampling date at the begin] Enrollment, First follow-up (Day 32), Fifth follow-up (1 year), Sixth follow-up (2 years)
  Palpate lymph nodes systematically, checking for size, consistency, mobility, and tenderness. Start with the cervical, axillary, and inguinal regions, then proceed to other areas if necessary. Normal lymph nodes should be small, mobile, and non-tender. Enlarged lymph nodes may suggest infection, inflammation, or malignancy. Assess their texture, whether soft or firm, and whether they are fixed or movable, as these characteristics can give clues about their underlying cause.
Spinal and Limb abnormalities in general physical condition as assessed by clinical examination | [set the tissue sampling date at the begin] Enrollment, First follow-up (Day 32), Fifth follow-up (1 year), Sixth follow-up (2 years)
  The examination is conducted according to the standards of the "Diagnostic Medicine (10th Edition, People's Medical Publishing House)".
  For the spine, observe posture and alignment, and palpate along the cervical, thoracic, and lumbar regions for tenderness, deformities, or abnormal curvatures. Test for flexibility by asking the patient to bend, twist, or rotate the spine. For the limbs, inspect the joints and muscles for symmetry, swelling, or signs of injury. Palpate for warmth, tenderness, or deformities in the joints. Assess the range of motion in both upper and lower limbs, testing for strength, coordination, and any signs of weakness or numbness.
Abdominal abnormalities in general physical condition as assessed by clinical examination | [set the tissue sampling date at the begin] Enrollment, First follow-up (Day 32), Fifth follow-up (1 year), Sixth follow-up (2 years)
  The examination is conducted according to the standards of the "Diagnostic Medicine (10th Edition, People's Medical Publishing House)".
  The abdominal examination involves inspection, palpation, percussion, and auscultation. Start by observing the abdomen for signs of distension, scars, or abnormalities in contour. Palpate gently for tenderness, masses, or organ enlargement. Percuss to assess for fluid buildup or gas, and auscultate for bowel sounds. Pay attention to any signs of pain during palpation, particularly in the liver, spleen, or lower abdomen, which may indicate underlying pathology such as infections, tumors, or gastrointestinal issues.
Neurological abnormalities in general physical condition as assessed by clinical examination | [set the tissue sampling date at the begin] Enrollment, First follow-up (Day 32), Fifth follow-up (1 year), Sixth follow-up (2 years)
  The examination is conducted according to the standards of the "Diagnostic Medicine (10th Edition, People's Medical Publishing House)".
  The neurological examination includes evaluating the patient's mental status, motor skills, coordination, and reflexes. Assess for any signs of cognitive impairment, speech difficulties, or mood changes. Test cranial nerve function, including vision, facial sensation, and strength. Evaluate motor function by observing muscle strength and tone, and test for signs of weakness or atrophy. Assess coordination with tasks such as finger-to-nose or heel-to-shin. Check for sensation abnormalities and perform reflex tests to assess the integrity of the central and peripheral nervous system.
Skin abnormalities in general physical condition as assessed by clinical examination | [set the tissue sampling date at the begin] Enrollment, First follow-up (Day 32), Fifth follow-up (1 year), Sixth follow-up (2 years)
  The examination is conducted according to the standards of the "Diagnostic Medicine (10th Edition, People's Medical Publishing House)".
  Examine the skin for color, texture, and any visible lesions, rashes, or scars. Look for signs of infection, redness, or swelling, and assess any pigmented lesions for irregularities in size, shape, or borders. Palpate the skin to check for moisture, temperature, and texture, noting any dryness, oiliness, or abnormalities. Inspect nails and hair for signs of systemic conditions. Look for bruising, ulcers, or signs of poor circulation, such as swelling or color changes in the extremities. The examination should also include a check for edema, especially in the lower limbs.

IPD SHARING:
Plan to Share IPD: No